CLINICAL TRIAL: NCT00361504
Title: A One-Year, Randomized, Open-Label, Parallel-Arm, Phase 3 Long-Term Safety Trial, With Controlled Adjustment of Dose, of Multiple Doses of CG5503 PR and Oxycodone CR in Subjects With Chronic Pain
Brief Title: A Study to Evaluate Long-Term Safety of Multiple Doses of Tapentadol (CG5503) Prolonged-Release (PR) and Oxycodone Controlled-Release (CR) in Patients With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR011074; R331333PAI3007 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee; Lower Back Pain; Pain
Keywords: Osteoarthritis; Pain; Low Back Pain; Hip Pain; Knee Pain; Backache; Tapentadol
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Low Back Pain; Pain; Osteoarthritis; Back Pain | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol (CG5503) (Experimental): Tapentadol (CG5503) extended release (ER) 100 to 250 mg twice daily (BID) for up to one year.
  Interventions: Drug: Tapentadol (CG5503) ER
- Oxycodone (Active Comparator): Oxycodone controlled release (CR) 20 to 50 mg twice daily (BID) for up to one year.
  Interventions: Drug: Oxycodone CR

INTERVENTIONS:
Drug: Oxycodone CR — Oxycodone CR 10 mg oral tablet BID administered for first 3 days, 20 mg oral tablet BID administered for next 4 days, 20 to 50 mg oral tablet BID administered for the next 51 weeks.
  Arms: Oxycodone
Drug: Tapentadol (CG5503) ER — Tapentadol (CG5503) ER 50 mg oral tablet BID administered for first 3 days, 100 mg oral tablet BID administered for next 4 days, 100 to 250 mg oral tablet BID administered for the next 51 weeks.
  Other Names: CG5503
  Arms: Tapentadol (CG5503)

SUMMARY:
The purpose of this study is to evaluate the safety profile of tapentadol (CG5503) PR at doses of 100 mg - 250 mg administered twice daily over a maximum one year period to patients with at least a 3-month history of low back pain, or pain caused by knee or hip osteoarthritis.

DETAILED DESCRIPTION:
Tapentadol (CG5503) is a centrally active pain-relieving drug being investigated for the treatment of acute and chronic pain. This study is a randomized (patients are assigned different treatments based on chance in a ratio of 4 patients on tapentadol (CG5503) PR to every 1 patient on oxycodone CR), open-label (both the Investigator and the patient know what medication is allocated), active-controlled, parallel-group, multicenter study. It is designed to investigate the long-term safety (side effects during up to one year of administration) and effectiveness (level of pain control) of tapentadol (CG5503) PR compared to oxycodone CR (an opioid commonly used for relief of moderate to severe pain) taken orally. The study consisted of a screening period (up to 14 days), a washout period (3 to 7 days), and an active treatment phase with titration and maintenance (total duration of 52 weeks). The doses of both of these medications will be adjusted to give the best therapeutic benefit for the patient. A total of 1123 patients will be screened. Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. Assessments of pain relief include the pain intensity numerical rating scale, and patient global impression of change scale (PGIC). Venous blood samples will be collected for the determination of serum concentrations of tapentadol (CG5503) and oxycodone. Tapentadol (CG5503) PR is also referred to as Tapentadol (CG5503) Extended Release (ER). Starting oral dose is randomly assigned to tapentadol (CG5503) PR 50 mg or oxycodone CR 10 mg twice daily (BID) x 3 days; then increase to tapentadol (CG5503)100 mg BID, oxycodone CR 20 mg BID x 4 days; during the maintenance phase upward titration may occur at a minimum of 3 day intervals in increments of tapentadol (CG5503) PR 50 mg BID or oxycodone CR 10 mg BID. The maximum doses are tapentadol (CG5503) PR 250 mg BID or oxycodone CR 50 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee or hip osteoarthritis with history of pain at the reference joint for at least 3 months or clinical diagnosis of low back pain of benign origin for at least 3 months
* Must be dissatisfied with their current analgesic therapy (e.g. Non-steroidal anti-inflammatory drugs NSAIDS, COX-2 inhibitors, opioids, paracetamol/acetaminophen
* Have a pain intensity >4 on Numerical Rating Scale

Exclusion Criteria:

* Life-long history of seizure disorder or epilepsy
* Any of the following within one year: mild/moderate traumatic brain injury, stroke, transient ischemic attack, and brain neoplasm
* Severe traumatic brain injury within 15 years (consisting of more than one of the following: brain contusion (injuries resulting in hemorrhage), intracranial hematoma, unconsciousness or post traumatic amnesia lasting for more than 24 hours) or residual sequelae suggesting transient changes in consciousness
* History of malignancy within past 2 years, with exception of a successfully treated basal cell carcinoma
* Presence of significant pain associated with conditions other than osteoarthritis or low back pain that could confound the assessment or self-evaluation of pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1123 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (52):
- United States (40):
  - Mesa, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Cudahy, California
  - Encinitas, California
  - San Diego, California
  - Westlake Village, California
  - Trumbull, Connecticut
  - Chiefland, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Oldsmar, Florida
  - Atlanta, Georgia
  - Cumming, Georgia
  - Decatur, Georgia
  - Perry, Georgia
  - Suwanee, Georgia
  - Woodstock, Georgia
  - Indianapolis, Indiana
  - Prairie Village, Kansas
  - Topeka, Kansas
  - Paducah, Kentucky
  - Baton Rouge, Louisiana
  - Rockville, Maryland
  - Wellesley Hills, Massachusetts
  - Kalamazoo, Michigan
  - Las Vegas, Nevada
  - Mamaroneck, New York
  - Williamsville, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Medford, Oregon
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Roanoke, Virginia
- Canada (12):
  - Edmonton, Alberta
  - Coquitlam, British Columbia
  - Halifax, Nova Scotia
  - Corunna, Ontario
  - Greater Sudbury, Ontario
  - Mississauga, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Vancouver, Ontario
  - Pointe-Claire, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Etropolski M, Kuperwasser B, Flugel M, Haufel T, Lange B, Rauschkolb C, Laschewski F. Safety and tolerability of tapentadol extended release in moderate to severe chronic osteoarthritis or low back pain management: pooled analysis of randomized controlled trials. Adv Ther. 2014 Jun;31(6):604-20. doi: 10.1007/s12325-014-0128-6. Epub 2014 Jul 2. PMID 24985410
- [Derived] Afilalo M, Morlion B. Efficacy of tapentadol ER for managing moderate to severe chronic pain. Pain Physician. 2013 Jan;16(1):27-40. PMID 23340531
- [Derived] Wild JE, Grond S, Kuperwasser B, Gilbert J, McCann B, Lange B, Steup A, Haufel T, Etropolski MS, Rauschkolb C, Lange R. Long-term safety and tolerability of tapentadol extended release for the management of chronic low back pain or osteoarthritis pain. Pain Pract. 2010 Sep-Oct;10(5):416-27. doi: 10.1111/j.1533-2500.2010.00397.x. PMID 20602712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this out-patient, multicenter study occurred between 14 November 2006 & 25 July 2008.
Pre-assignment Details: In this study 1123 participants passed screening, 1121 participants were randomized (2 participants were not randomized in error) & 1117 participants received at least 1 dose of study medication (4 participants did not receive study medication)
Period: Overall Study
Arm/Group | Tapentadol (CG5503) | Oxycodone
Started | 894 (Number of participants who received at least 1 dose of study medication) | 223 (Number of participants who received at least 1 dose of study medication)
Completed | 413 | 78
Not Completed | 481 | 145
Not completed — Withdrawal by Subject | 94 | 31
Not completed — Lost to Follow-up | 40 | 7
Not completed — Adverse Event | 203 | 82
Not completed — Lack of Efficacy | 72 | 7
Not completed — Resolution of Pain | 2 | 0
Not completed — Study medication non compliant | 42 | 15
Not completed — All other | 28 | 3

BASELINE CHARACTERISTICS:
Groups:
- Tapentadol (CG5503): Tapentadol (CG5503) extended release (ER) 100 to 250mg twice daily (BID) for up to one year
- Oxycodone: Oxycodone controlled release (CR) 20 to 50mg twice daily (BID) for up to one year.
- Total: Total of all reporting groups
Arm/Group | Tapentadol (CG5503) | Oxycodone | Total
Number analyzed (Participants) | 894 | 223 | 1117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 649 | 156 | 805
  >=65 years | 245 | 67 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.51) | 58.1 (11.83) | 57.0 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 515 | 125 | 640
  Male | 379 | 98 | 477
Region of Enrollment [Number; unit: participants]
  North America | 684 | 170 | 854
  Europe | 210 | 53 | 263

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: The number of participants who reported a TEAE during the treatment period. TEAE was defined as any adverse event that started or worsened on or after the start of the study medication and up to 3 days after the discontinuation of the study medication.
Time Frame: 52 weeks
Population: Safety analysis set (All randomized participants who took at least one dose of study medication).
Measure: Number; unit: Participants
Arm/Group | Tapentadol (CG5503) | Oxycodone
Number analyzed (Participants) | 894 | 223
Participants | 766 (2.986) | 202 (2.470)

2. Secondary Outcome: Change From Baseline in Average Pain Intensity Scores at Week 52 Using the Numerical Rating Scale (NRS)
Description: The Participants indicated the average level of pain experienced, at each study visit, over the previous 24 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". Baseline was the average pain intensity scores measured prior to randomization (At Week 1). At Week 52 again the average pain intensity scores were collected and the change in scores at Week 52 from the baseline scores was considered as the change from baseline in average pain intensity scores at Week 52.
Time Frame: Baseline, Week 52
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Tapentadol (CG5503) | Oxycodone
Number analyzed (Participants) | 821 | 178
Scores on a Scale | -3.22 (2.664) | -3.14 (2.409)

ADVERSE EVENTS:
Arm/Group | Tapentadol (CG5503) | Oxycodone
Serious Adverse Events (participants affected / at risk) | 49/894 | 9/223
Other Adverse Events (participants affected / at risk) | 766/894 | 202/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (CG5503) (N=894) | Oxycodone (N=223)
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0
Colonic Polyp (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diabetic Gastroparesis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Drug Withdrawal Syndrome (General disorders) | 1 | 0
Hernia Obstructive (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Treatment Failure (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Nerve Compression (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Euphoric Mood (Psychiatric disorders) | 1 | 0
Substance Abuse (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyoid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Visual Disturbance (Eye disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Breast Mass (Reproductive system and breast disorders) | 1 | 0
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (CG5503) (N=894) | Oxycodone (N=223)
Constipation (Gastrointestinal disorders) | 202 | 86
Nausea (Gastrointestinal disorders) | 162 | 74
Dry Mouth (Gastrointestinal disorders) | 81 | 10
Diarrhoea (Gastrointestinal disorders) | 71 | 12
Vomiting (Gastrointestinal disorders) | 63 | 30
Somnolence (Nervous system disorders) | 133 | 25
Dizziness (Nervous system disorders) | 132 | 43
Headache (Nervous system disorders) | 119 | 17
Nasopharyngitis (Infections and infestations) | 49 | 6
Sinusitis (Infections and infestations) | 33 | 13
Insomnia (Psychiatric disorders) | 60 | 9
Fatigue (General disorders) | 87 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 48 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less